CLINICAL TRIAL: NCT04333394
Title: Investigating the Effectiveness of Probiotic Supplement in Improving Attention Deficit Hyperactivity Disorder Symptoms in Children
Brief Title: Effectiveness of Probiotic Supplement In Improving Attention Deficit Hyperactivity Disorder Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 96/114
Record Dates: First submitted 2020-03-24; First posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD, Probiotics, Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The present study will be conducted as a phase 3, randomized double-blind placebo-controlled trial on 40 attention deficit hyperactivity disorder patients allocated in 2 parallel groups each consisted of 20 patients who will receive Probiotic or placebo. From the beginning of the study, A and B codes are available to researchers to recruit the patients using ten 4-Block Randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both patients and researchers won't be aware of the treatments patients receiving in this study (unaware of the quiddity of A and B capsules), so the study has a double-blind design. Only one of the staff of the company that supplied the Probiotic supplement is aware of the type of assigned intervention for each patient. After collecting the data, he will unseal the codes for researchers, the statistical analyst, participants and those who prepare the manuscript.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Active Comparator): The probiotics capsules contain 7 strains of friendly bacteria (Lactobacillus casei PXN 37, Lactobacillus rhamnosus PXN 54, Streptococcus thermophilus PXN 66, Bifidobacterium breve PXN 25, Lactobacillus acidophilus PXN 35, Bifidobacterium longum PXN 30, Lactobacillus bulgaricus PXN 39)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo capsules have an identical appearance to probiotic capsules and contain microcrystal cellulose.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic capsules will be administrated once a day. medication with Ritalin starts at the onset of the study in a dose-dependent manner and simultaneous with probiotic supplementation.
  Arms: Probiotic
Other: Placebo — The placebo capsules will be administered once a day. medication with Ritalin starts at the onset of the study in a dose-dependent manner and simultaneous with placebo supplementation.
  Arms: Placebo

SUMMARY:
To study the effects of probiotic supplement in children with Attention-deficit hyperactivity disorder (ADHD),40 patients will be randomly allocated to two groups of intervention and placebo. The intervention and the placebo group will be prescribed with 1 capsule of probiotics and placebo for 8 weeks, respectively. Treatment efficacy will be assessed via administrating the Conners's rating

DETAILED DESCRIPTION:
Both probiotics and placebo groups will receive medication with Ritalin in a dose-dependent manner, starting at the onset of the study and simultaneous with probiotic supplementation. Children weighed 30 Kg or less receive 0.3 mg/kg of Ritalin in 3 separate intervals and after four weeks the dosage will increase to 0.5mg/kg. Those who weighed more than 30 kg receive 0.5 mg/kg with the same pattern that reaches the highest point of 0.7 mg/kg by week four. Each dosage will be administrated trice a day with breakfast, lunch, and dinner. In the middle of the study patients who consumes less than 80% of their supplements will be omitted from the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Attention Deficit Hyperactivity Disorder
* Having an Intelligence quotient more than 85 based on Wechsler test for children
* Willing to participate in the study

Exclusion Criteria:

* History of any other mental and psychological disorder such as depression, chronic motor tic disorder, communication disorder, learning disability
* Taking any stimulant, sedative, anti-anxiety and anti-psychotic medications
* History of any chronic disorders, requiring long term medication (such as cancers, Cirrhosis, autoimmune disorders, metabolic disorders ) or, chronic neurological disorders (such as epilepsy)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
symptoms of Attention-deficit hyperactivity disorder (ADHD) | 8 weeks
  symptoms were assessed using Conners's scale
The severity of the Attention-deficit hyperactivity disorder (ADHD) | 8 weeks
  The severity of the ADHD was assessed using the Clinical Global Impression (CGI) test

CONTACTS AND LOCATIONS:
Overall Officials: Soodeh Razeghi Jahromi, PhD, Study Director — Shahid Beheshti University of Medical Sciences
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehrān, Tehran Province, Iran